CLINICAL TRIAL: NCT01748214
Title: Premature Infant Exposure to Noise Generated by Respiratory Support
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jonathan Swanson, MD, Prinicipal Investigator, University of Virginia
Other Study IDs: 13164
Record Dates: First submitted 2012-12-06; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Premature Birth of Newborn
Keywords: continuous positive airway pressure; high flow nasal cannula; hearing outcomes; noise exposure; preterm infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nasal CPAP: Infants received nasal CPAP as standard of care.
- High Flow Nasal Cannual: Infants received high flow nasal cannula as standard of care.

SUMMARY:
Infants in neonatal intensive care units are increasing exposed to non-invasive ventilatory support modes (nasal continuous positive airway pressure - NCPAP and high flow nasal cannula: >1 L/min flow - HFNC). While there have been small descriptive studies of noise exposure in infants on NCPAP, there have been no comparative trials done comparing noise exposure in infants undergoing both NCPAP and HFNC.

Objective: Using a cross-over model determine noise exposure levels in infants exposed to similar levels of respiratory support provided by NCPAP and HFNC.

DETAILED DESCRIPTION:
Infants born < 32 weeks, in an incubator, and > 7 days postnatal that were maintained on either on NCPAP or HFNC to maintain SaO2 in a range of 88 - 92 %. Study infants had decibel measurements obtained every 15 seconds for 30 minutes using a noise dosimeter (NoisePro DLX-1). The microphone for the dosimeter was suspended from the inside of the incubator such that it hung 1 foot above the infants nose and mouth. The exhalation port for NCPAP was placed outside of the incubator. Repeated measurement periods on the same mode of support were made within a 72 hour period. Each infant the acted as their own control and was switched within 7 days to the alternative respiratory support method that maintained similar SaO2 goals and repeat measurements were obtained. Comparisons of mean decibel levels during recording were compared using paired t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant born < 32 weeks and 0 days post-conceptional age;
* Seven or more days of age and not in acute respiratory distress;
* Need for nasal continuous positive airway pressure or high-flow nasal cannula for ventilation or supplemental oxygen delivery;
* In a neutral-thermal environment (i.e. isolette)

Exclusion Criteria:

* Oro-facial congenital anomalies;
* Congenital heart disease (except for patent ductus arteriosus and/or patent foramen ovale);
* Unstable respiratory status as deemed by the attending physician
* Patients under isolation for infectious disease

Min Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born < 32 weeks, in an incubator, and > 7 days postnatal admitted to the Newborn Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Noise level | 6 days
  Noise levels will be measured during a set time while infants are on Nasal CPAP and Nasal High flow cannula as standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Attridge, MD, Principal Investigator — UVA School of Medicine
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States